CLINICAL TRIAL: NCT01229917
Title: Rhinovirus Study With Lactobacillus Rhamnosus GG
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Valio Ltd (Industry)
Collaborators: University of Helsinki (Other); University of Virginia (Other); Medcare Ltd (Unknown)
Other Study IDs: Valio-73
Record Dates: First submitted 2010-10-26; First posted 2010-10-28 (Estimated); Last update posted 2011-07-07 (Estimated); Status verified 2011-07

CONDITIONS: Respiratory Tract Infections [C08.730]
MeSH Terms: interventions — Fruit and Vegetable Juices

INTERVENTIONS:
Other: Fruit juice with Lactobacillus rhamnosus GG, version 1
Other: Fruit juice with Lactobacillus rhamnosus GG, version 2
Other: Standard fruit juice

SUMMARY:
The purpose of this study is to evaluate the symptom impact of probiotic Lactobacillus rhamnosus GG during rhinovirus infection.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female in general good health (stabilized chronic illnesses and regular medications are accepted, if not otherwise mentioned in the exclusion criteria)
2. Age 18-65 years
3. Serum neutralizing antibody titer of 1:4 or less for the challenge rhinovirus
4. No clinically significant finding on the pre-study nasal examination
5. Females must have a negative urine pregnancy test, and women of child-bearing potential must be using an effective method of birth control such as, but not limited to birth control pills, contraceptive foam, diaphragm, IUD, surgical sterilization, abstinence, or condoms
6. Written informed consent must be obtained at enrollment into the study

Exclusion Criteria:

1. Suffer from or have a history of significant allergic rhinitis at the time of study
2. Bronchial asthma or other lower respiratory tract diseases, such as chronic obstructive lung disease or emphysema
3. Nasal abnormalities or other nasal pathology, such as irreversible nasal mucosal hypertrophy or severe nasal septum derivation
4. Pregnancy or lactation
5. History of alcohol abuse (regularly consumes 5 or more alcohol drinks per day) and/or drug abuse during the 12 month period immediately preceding study enrollment
6. Daily smoking within the past 2 years
7. Use of investigational product or participation in a device trial during the 30 day period immediately preceding study enrollment
8. Previous participation in an experimental study with rhinovirus 39
9. Allergy to any ingredient in the study product
10. Have, as determined by the investigator and/or the sponsor's medical monitor, any surgical or medical condition or take any medication or dietary supplement that could interfere with the interpretation of study results or jeopardize the safety of the subject

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Birgit Winther, Dr., Principal Investigator — University of Virginia Health System
Locations (1):
- University of Virginia, Respiratory Disease Study Center, Charlottesville, Virginia, United States